CLINICAL TRIAL: NCT06572644
Title: Evaluation of a Highly Sensitive Rapid Diagnostic Test for Detecting Falciparum Malaria Infection in Pregnancy in Burkina Faso
Brief Title: Performance of an Ultrasensible Malaria Rapid Diagnostic Test Among Pregnant Women in Burkina Faso
Acronym: HS-RDT-MiP
Status: Completed | Type: Observational
Sponsor: Centre MURAZ/Institut National de Santé Publique (Other Government)
Collaborators: University of Ghana (Other)
Responsible Party: Principal Investigator, Mamoudou Cissé, Assistant Professor of Parasitology and Mycology, Centre MURAZ/Institut National de Santé Publique
Other Study IDs: INSP_CM_09_2022
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Malaria,Falciparum
Keywords: Pregnancy; Malaria; Performance; Ultrasensible rapid diagnostic test; Burkina Faso
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Dried blood spots were collected at enrolment and one month after sulfadoxine-pyrimethamine uptake.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the diagnostic performance of the highly sensitive rapid diagnostic test (HS-RDT) compared to an ultrasensitive qPCR for detection of falciparum malaria in pregnant women attending antenal care (ANC) in Burkina Faso. The main question it aims to answer is:

• What are the sensitivity and specificity of the HS-RDT compared to ultrasensitive quantitative polymerase chain reaction (qPCR) considered as gold standard for dection of falciparum malaria in pregnant women attending ANC in Burkina Faso ? Participants will be included during their ANC visits and screened for malaria using the HS_RDT, the conventional RDT (Co_RDT), microscopy, and qPCR.

DETAILED DESCRIPTION:
A cross-sectional study including 288 pregnant women was conducted at the Centre médical urbain (CMU) of Lafiabougou located in the periurban area of Bobo-Dioulasso the second largest city of Burkina Faso. Pregnant women attending their ANC visits at the CMU of Lafiabougou were recruited and enrolled into the study if eligible criteria were fulfilled.

At enrolment, an individual structured questionnaire was administered to the selected pregnant women and their sociodemographic data (age, educational level, and profession) and history of illness was collected. In addition, obstetric history (parity, gestational age, number of ANC visits, uptake of IPTp-SP) and clinical information (body temperature, weight, height, and arm circumference) were recorded. Thereafter, a venous blood sample (5 mL) was collected to screen for malaria infection (based on HS-RDT, Co_RDT, and thick and thin blood smears), dried blood spots (DBS) (for molecular studies), and haemoglobin concentration measurement. The remaining blood sample was stored for future studies.

After enrolment, only pregnant women eligible for their first IPTp-SP dose uptake was followed up for 30 days to assess the impact of IPTp-SP on both falciparum parasitaemia and falciparum resistant strains. At the end of follow up, a venous blood sample (5 mL) was collected for thick and thin blood smears, DBS, and haemoglobin concentration measurement. The remaining blood sample was stored for future studies.

All biological samples was collected and stored at ambient temperature before being transported to the Laboratory of Parasitology of Centre MURAZ and processed.

The index tests included HS_RDT (NxTek Eliminate Malaria Pf, product code 05FK140, batch No. 05LDG008B, Alere/Abbott, Republic of Korea), Co_RDT (AdvDxTM Malaria Pf, product code 004ADFEF025KI-2, batch No. ADF77/0222, Advy Chemical, India), and light microscopy.

The ultrasensitive qPCR assay targeting the multicopy conserved var gene acidic terminal sequence (varATS) (Hofmann et al. 2015) was used as gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Living in Bobo-Dioulasso for at least 6 months before the beginning of the study ;
* Provision of informed consent.

Exclusion Criteria:

* Past history of malaria or antimalarial drugs within the last 3 months ;
* Having tested positive for malaria by microscopy or RDT in any previous ANC visit ;
* Symptoms and signs of severe malaria as defined by WHO.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women attending their ANC visits at the Centre Médical Urbain de Lafiabougou
Sampling Method: Probability Sample
Enrollment: 288 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity of HS_RDT | At baseline
  It is defined as the proportion of positives that are correctly identified when compared with the gold standard (qPCR).
Specificity of HS_RDT | At baseline
  It is defined as proportion of negatives that are correctly identified when compared with the gold standard (qPCR).

SECONDARY OUTCOMES:
Positive predictive value | At baseline
  Probability that P. falciparum infection is present when HS_RDT, Co_RDT, and microscopy are positive
Negative predictive value | At baseline
  Probability that P. falciparum infection is not present when HS_RDT, Co_RDT, and microscopy are negative
The prevalence of Pfhrp2 and Pfhrp3 genes deletions among the study participants | At baseline
  Proportion of pregnant women with malaria parasites carrying Pfhrp2/Pfhrp3 deletions
Impact of intermittent preventive treatment in pregnancy with sulfadoxine-pyrimethamine (IPTp- SP) on falciparum parasitaemia | 30 days after uptake of IPTp-SP
  Proportion of pregnant women with falciparum parasitaemia 30 days after uptake of IPTp-SP

OTHER OUTCOMES:
Prevalence of anaemia | At baseline
  Proportion of pregnant women with haemoglobin concentration <11 g/dL
Prevalence of Pfdhfr & Pfhdps mutations | At baseline
  Proportion of pregnant women with Pfdhfr (N51I, C59R, S108N, I164L) and Pfdhps (A437G, K540E) mutations

CONTACTS AND LOCATIONS:
Overall Officials: Mamoudou Cissé, MD, PhD, Principal Investigator — Centre MURAZ/Institut National de Santé Publique
Locations (1):
- Centre Médical Urbain de Lafiabougou, Bobo-Dioulasso, Houet, Burkina Faso